CLINICAL TRIAL: NCT00909181
Title: A Double-Blind, Randomized, Parallel, Placebo-Controlled, Multicenter Study Evaluating the Effect of Treatment With Topically Administered Oxybutynin Gel in Patients With Urinary Frequency, and Urge and Mixed Urinary Incontinence With a Predominance of Urge Incontinence Episodes With an Open-Label Extension
Brief Title: Study of Topically Administered Oxybutynin Gel in Patients With Urge Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Antares Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20070060
Record Dates: First submitted 2009-05-25; First posted 2009-05-27 (Estimated); Results first posted 2011-01-19 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Urge Urinary Incontinence; Urinary Frequency
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — oxybutynin; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oxybutynin Gel 56 mg/day (Experimental)
  Interventions: Drug: Oxybutynin; Drug: Placebo
- Oxybutynin Gel 84 mg/day (Experimental)
  Interventions: Drug: Oxybutynin; Drug: Placebo
- Placebo Gel (Placebo Comparator)
  Interventions: Drug: Oxybutynin; Drug: Placebo

INTERVENTIONS:
Drug: Oxybutynin — Oxybutynin Gel. Transdermal gel was applied once-daily (in the morning) during 12 weeks of treatment.
  Evaluation: reduction of incontinent episodes (baseline vs 12 weeks); comparison 56 resp. 84 mg vs placebo
  Other Names: Anturol; Oxybutynin Gel 3%
Drug: Placebo — Placebo Gel Oxybutynin Gel. Transdermal gel was applied once-daily (in the morning) during 12 weeks of treatment.
  Evaluation: reduction of incontinent episodes (baseline vs 12 weeks); comparison 56 resp. 84 mg vs placebo
  Other Names: Anturol; Oxybutynin Gel 3%

SUMMARY:
The primary objective of the double-blind phase of the study is to compare the effects of two doses of oxybutynin gel to placebo gel. The objective of the open-label extension is to evaluate the extended safety and skin-irritation profile of topically administered oxybutynin gel.

The hypothesis is that topically administered oxybutynin gel will decrease (compared to placebo) the number of incontinence episodes per week, average daily urinary frequency, and urinary urgency; increase average urinary void volume; and improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Overactive bladder (OAB) symptoms of urge and/or mixed UI with a predominance of urge incontinence for at least 3 months
* Have a history of at least 1 - 2 urge episodes and 8 or more voids per day

Exclusion Criteria:

* Incontinence that is predominantly stress, insensate, or overflow in nature, or incontinence related to chronic illness, anatomical weakness/abnormalities or concomitant medications
* PVR volume > 200 mL or relative PVR > 50% of pre-void volume as determined by bladder ultrasound
* History of urinary retention, gastric retention, or uncontrollable narrow-angle glaucoma, or patients who are at risk for these conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (53):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Laguna Hills, California
  - Los Angeles, California
  - San Diego, California
  - Farmington, Connecticut
  - New Britain, Connecticut
  - New Port Richey, Florida
  - North Miami, Florida
  - Pembroke Pines, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Columbus, Georgia
  - Sandy Springs, Georgia
  - Stockbridge, Georgia
  - Evanston, Illinois
  - West Des Moines, Iowa
  - Shreveport, Louisiana
  - Annapolis, Maryland
  - Towson, Maryland
  - Watertown, Massachusetts
  - Grand Rapids, Michigan
  - Saginaw, Michigan
  - Chesterfield, Missouri
  - Las Vegas, Nevada
  - Brooklyn, New York
  - Endwell, New York
  - Kingston, New York
  - Poughkeepsie, New York
  - Williamsville, New York
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Harrisburg, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Wadsworth, Ohio
  - Bethany, Oklahoma
  - Corvallis, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Landsdale, Pennsylvania
  - Greenville, South Carolina
  - Mt. Pleasant, South Carolina
  - Myrtle Beach, South Carolina
  - Sioux Falls, South Dakota
  - Fayetteville, Tennessee
  - Provo, Utah
  - Richmond, Virginia
  - Seattle, Washington
  - Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in clinical sites (urologists mainly) started in September 2007 and was terminated in February 2010.
Pre-assignment Details: Baseline period was 1 week. Patients on OAB drugs had to wash out.
Period: Overall Study
Arm/Group | Oxybutynin Gel 56 mg/Day | Oxybutynin Gel 84 mg/Day | Placebo Gel
Started | 210 | 214 | 202
Completed | 171 | 196 | 169
Not Completed | 39 | 18 | 33
Not completed — Lost to Follow-up | 39 | 18 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxybutynin Gel 56 mg/Day | Oxybutynin Gel 84 mg/Day | Placebo Gel | Total
Number analyzed (Participants) | 210 | 214 | 202 | 626
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 120 | 122 | 120 | 362
  >=65 years | 90 | 92 | 82 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (12.6) | 59.1 (13.3) | 57.8 (13.3) | 58.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 182 | 178 | 542
  Male | 28 | 32 | 24 | 84
Region of Enrollment [Number; unit: participants]
  United States | 210 | 214 | 202 | 626
Number of incontinent episodes at baseline [Mean (Standard Deviation); unit: Episodes] | 50.1 (32.5) | 43.6 (27.5) | 45.8 (28.9) | 46.5 (29.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Weekly Frequency of Urinary Incontinence Episodes at Week 12
Description: Reduction in number of incontinent episodes, evaluated as mITT (modified intention to treat), after 12 weeks of treatment compared to baseline.
Time Frame: 12 weeks
Population: mITT (modified intended to treatment) per protocol Difference between Baseline and after 12 weeks treatment
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Oxybutynin Gel 56 mg/Day | Oxybutynin Gel 84 mg/Day | Placebo Gel
Number analyzed (Participants) | 175 | 191 | 166
Episodes | -24.8 (28.7) | -21.9 (25.1) | -20.0 (27.0)

ADVERSE EVENTS:
Time Frame: Throughout whole study (20 months)
Arm/Group | Oxybutynin Gel 56 mg/Day | Oxybutynin Gel 84 mg/Day | Placebo Gel
Serious Adverse Events (participants affected / at risk) | 3/210 | 4/214 | 2/202
Other Adverse Events (participants affected / at risk) | 98/210 | 90/214 | 53/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxybutynin Gel 56 mg/Day (N=210) | Oxybutynin Gel 84 mg/Day (N=214) | Placebo Gel (N=202)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion missed (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hepatic neoplasm malignant (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxybutynin Gel 56 mg/Day (N=210) | Oxybutynin Gel 84 mg/Day (N=214) | Placebo Gel (N=202)
Dry mouth (Gastrointestinal disorders) | 23 | 26 | 10
Constipation (Gastrointestinal disorders) | 3 | 8 | 5
Diarrhoe (Gastrointestinal disorders) | 5 | 2 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 10
Urinary tract infection (Infections and infestations) | 9 | 6 | 4
Nasopharyngitis (Infections and infestations) | 5 | 5 | 0
Sinusitis (Infections and infestations) | 5 | 3 | 2
Application site reaction (Skin and subcutaneous tissue disorders) | 5 | 3 | 0
Headache (Nervous system disorders) | 6 | 6 | 8
Dizziness (Nervous system disorders) | 6 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 5
Application site erythema (General disorders) | 8 | 8 | 2
Application site rash (General disorders) | 9 | 7 | 1
Application site pruritus (General disorders) | 3 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less